CLINICAL TRIAL: NCT01515410
Title: A Phase 2, Randomized, Open-Label, Crossover Study to Compare DM-1992, a Novel Gastric-Retentive Extended-Release Formulation of Levodopa/Carbidopa, to an Immediate-Release Carbidopa Tablet in Patients With Advanced Parkinson's Disease With Motor Fluctuations
Brief Title: Study in Advanced Parkinson's Disease Patients With Predictable Motor Fluctuations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Depomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 81-0068
Record Dates: First submitted 2012-01-11; First posted 2012-01-24 (Estimated); Results first posted 2014-03-10 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2012-11

CONDITIONS: Parkinson's Disease; Motor Fluctuations
Keywords: Parkinson's disease; PD; stage2/3Parkinson's; Advanced Parkinson's Disease with Motor Fluctuations
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DM-1992 (Experimental): DM-1992, a gastric-retentive extended-release tablet containing 72.5mg carbidopa (CD) and 230mg levodopa (LD)
  Interventions: Drug: DM-1992
- Sinemet IR (Active Comparator): An Immediate-release (IR) tablet containing 25mg carbidopa (CD) and 100mg levodopa (LD)
  Interventions: Drug: Sinemet IR

INTERVENTIONS:
Drug: DM-1992 — 72.5mg carbidopa/230mg levodopa
  Arms: DM-1992
Drug: Sinemet IR — Immediate-release tablet containing 25mg carbidopa and 100mg levodopa
  Arms: Sinemet IR

SUMMARY:
The primary objective of this study is to explore the efficacy and tolerability of DM-1992 compared to a standard carbidopa/Levodopa Immediate-Release (CD/LD IR) tablet (Sinemet IR) as measured by:

* "ON" time with no dyskinesia or non-troublesome dyskinesia
* "OFF" time

ELIGIBILITY:
Inclusion Criteria:

1. Men and women at least 30 years and older at the time of informed consent with advanced idiopathic Parkinson's disease with predictable wearing-off motor fluctuations with Hoehn and Yahr Stage II-III when "on."
2. Patients should be able to differentiate between the "ON" and "OFF" states with an average daily "OFF" time of ≥ 2.5 hours at study entry.
3. On a stable daily dose of LD of ≥ 400 mg but ≤1600 mg for at least 1 month prior to the screening visit.
4. Non CD/LD containing anti-Parkinson's medications should be kept at stable doses for 1 month prior to screening visit. Patients should be willing to keep their non LD containing medications consistently throughout the study duration.
5. Female patients of childbearing potential should be abstinent or continuing to practice and willing to continue throughout the study with appropriate contraceptives (defined as Nova ring, oral, injected, transdermal patch, implanted, or barrier).
6. Mini Mental State Examination (MMSE) ≥ 26 at screening visit.
7. Able to provide informed consent and willing to sign Health Insurance Portability and Accountability Act (HIPAA) authorization.
8. Able and willing to comply with the protocol, including availability for all scheduled study visits and blood sample collections. Must be under the observation of a competent care giver throughout the study participation.

Exclusion Criteria:

1. Patients with atypical or drug-induced Parkinson's disease.
2. Patients with a known history of hypersensitivity to levodopa or carbidopa.
3. Patients who receive treatments with dopamine receptor blocking agents
4. Patients with a history of seizures except of childhood febrile seizure.
5. Patients with dementia.
6. Patients with a significant history of GI diseases (severe inflammatory bowel disease, irritable bowel disease, dyspepsia, gastro-esophageal reflux disease etc.) in the past five years.
7. Patients with any history of gastric surgery other than vagotomy and pyloroplasty.
8. Patients with an immune-compromised state.
9. Patients with clinically significant hepatic insufficiency with Child-Pugh total score of ≥ 5.
10. Patients with a calculated creatinine clearance (Clcr) < 50 mL/min using the Cockcroft-Gault equation.
11. Patients who have a difficulty swallowing tablets.
12. Patient has participated in a clinical trial of an investigational drug or device within 30 days of the screening visit.
13. Patients with any other serious medical condition that, in the opinion of the Investigator would jeopardize the safety of the patient or affect the validity of the study results.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rekha Sathyanarayana, Study Director — Depomed
Locations (7):
- United States (7):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Long Beach, California
  - Chicago, Illinois
  - Bingham Farms, Michigan
  - Cincinnati, Ohio
  - Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 34 subjects were randomly assigned to treatment in this crossover study: 19 in the DM-1992 for Period 1 and Sinemet IR for Period 2 sequence, and 15 in the Sinemet IR for Period 1 and DM-1992 for Period 2 sequence. All 34 subjects received study treatment and were included in the safety and intent-to-treat (ITT) populations.
Groups:
- DM-1992 First, Then Sinemet IR: DM-1992, a gastric-retentive extended-release tablet containing 72.5mg carbidopa (CD) and 230mg levodopa (LD) first, then Sinemet IR, an Immediate-release (IR) tablet containing 25mg carbidopa (CD) and 100mg levodopa (LD)
- Sinemet IR First, Then DM-1992: Sinemet IR, an Immediate-release (IR) tablet containing 25mg carbidopa (CD) and 100mg levodopa (LD) first, then DM-1992, a gastric-retentive extended-release tablet containing 72.5mg carbidopa (CD) and 230mg levodopa (LD)
Period: Overall Study
Arm/Group | DM-1992 First, Then Sinemet IR | Sinemet IR First, Then DM-1992
Started | 19 | 15
Completed | 19 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: DM-1992 first, then Sinemet IR; Sinemet IR first, then DM-1992
Arm/Group | Overall Study
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (8.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 26
Race/Ethnicity, Customized [Number; unit: participants]
  White | 32
  Afro-Caribbean | 2
  Native Hawaiian or Other Pacific Islander | 0
  Asian | 0
  American Indian or Alaskan Native | 0
  Hispanic or Latino | 0
  Other | 0
Percent "OFF" Time (%) [Mean (Standard Deviation); unit: percentage of time] — Baseline is the average of the 3 days recorded in the patient diary prior to Day 1 of Period 1.
  percentage of time | 32.50 (9.962)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective of This Study is to Explore the Efficacy and Tolerability of DM-1992 Compared to a Standard CD/LD IR Formulation as Measured by Percent "OFF" Time.
Description: "OFF" indicates wearing off motor fluctuations before the next levodopa dose. Percent "OFF" time is calculated as the total "OFF" time divided by the total awake time for each day and multiplied by 100.
  Patient diary-every 30min while awake for 3days prior to initial Day1 as baseline & during the last 3days before Day10 for both treatments for dyskinesia state.
  Baseline is the average of the 3 days recorded in the patient diary prior to Day 1 of Period 1.
  End of Period is the average of the 3 days recorded in the patient diary prior to Day 10 in each period.
  Clinician-Assess efficacy at pre-dose, every 30min for Day1 and hourly for Day10 for dyskinesia state & motor fluctuations at clinic visits.
Time Frame: Baseline and 10 days for each of the 2 study periods
Population: Modified Intent-to-treat (ITT) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of time
Groups:
- Sinemet IR: Sinemet IR, an Immediate-release (IR) tablet containing 25mg carbidopa (CD) and 100mg levodopa (LD)
Arm/Group | DM-1992 | Sinemet IR
Number analyzed (Participants) | 34 | 34
percentage of time | -5.52 [-10.42 to -0.63] | 1.33 [-3.56 to 6.22]
Statistical Analysis 1: Comparison: DM-1992 vs Sinemet IR; Percent "OFF" Time (%); Test type: Superiority or Other; p = 0.0471, ANCOVA — This p-value indicates statistical significance at the 0.05 level; No subjects early-terminated from the study; Difference in Least Squares Mean = -6.86, 95% CI [-13.62 to -0.09]

ADVERSE EVENTS:
Time Frame: Adverse events collected for a total of 5-6 weeks: from after signing the informed consent to the end of the study (Period 2, Day 10).
Description: Adverse event collection began after signing the informed consent and continued through Period 2, Day 10; serious adverse events followed for 30 days after study completion.
Arm/Group | DM-1992 | Sinemet IR
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 12/34 | 4/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DM-1992 (N=34) | Sinemet IR (N=34)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Parkinsonian gait (Nervous system disorders) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Hypertonia (Nervous system disorders) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees that sponsor shall have the right to the first publication of the study results which is intended to be a joint, multi-center publication. Following the first publication, the PI may publish study data or results, provided however PI submits the proposed publication to sponsor for review at least 60 days prior to the date of the proposed publication. Sponsor may remove any information that is considered confidential and/or proprietary other than study data.